CLINICAL TRIAL: NCT06625762
Title: Nantes Bariatric Surgery Cohort
Acronym: NBC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC23_0004
Record Dates: First submitted 2024-09-03; First posted 2024-10-03 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-06

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Biological aging; Adipocyte dysfunction; Biological rhythms
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- observation of the change in biological age after bariatric surgery (Other): Patients over 18 years of age suffering from obesity and requiring bariatric surgery.
  Evolution of biological age 1 year after surgery, defined by the difference between age biological at TPO and TAC 1 year, estimated by measuring the phenotypic age, itself determined from the following eight variables: albumin; creatinine; fasting blood sugar; CRP
  ; lymphocyte count; mean corpuscular volume of red blood cells; Anisocytosis index of red blood cells; alkaline phosphatases; leukocyte rate.
  Interventions: Other: Nantes bariatric surgery cohort

INTERVENTIONS:
Other: Nantes bariatric surgery cohort — The participants will be individuals living with obesity undergoing bariatric surgery

SUMMARY:
While current research suggests that inflammation of adipose tissue in obesity is linked to accelerated aging, it has yet to be determined in humans how this could enhance preventative and personalized medicine for obese individuals. The NBC study aims to investigate :

1. Whether bariatric surgery is associated with changes in biological age
2. If bariatric surgery alters adipocyte dysfunction, the microbiota and biological rhythms
3. Whether changes in adipocyte dysfunction, microbiota and biological rhythms are linked to changes in biological age.

To achieve this, establishing a biocollection before, during and after bariatric surgery will be crucial in addressing these questions

DETAILED DESCRIPTION:
The study of the Nantes Bariatric Surgery Cohort (NBC) aims to evaluate the impact of bariatric surgery on biological age, adipocyte dysfunction, microbiota, and biological rhythms in individuals with obesity. This observational study will include 300 participants over 3.5 years. It involves pre-operative, peri-operative, and post-operative visits to collect clinical, biological, and lifestyle data. Key assessments include anthropometrics, blood tests, questionnaires, and biocollections

ELIGIBILITY:
Inclusion Criteria :

Individuals selected for bariatric surgery (starting the BC pathway within the Nantes University Hospital bariatric unit). Inclusion criteria are those of the Bariatric Surgery program.

* male or female, adult over 18 years of age
* BMI ≥ 35 kg/m2 with complication(s) or ≥ 40 kg/m2 with or without complication (the list of eligible complications is referenced in HAS 2024 recommendations). In the event of a change in access to bariatric surgery, this threshold could be revised without any substantial change to the protocol.
* having consented to their participation in the cohort
* participant affiliated to or benefiting from a social security scheme

Exclusion Criteria :

* Persons protected by law (guardianship or trusteeship) or deprived of their freedom,
* Pregnant women (contraindication to CB) or nursing mothers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Observe how biological age evolves between pre-bariatric surgery and 1 year after bariatric surgery | 1 year
  Biological age will be estimated by measuring phenotypic age. The phenotypic age will be determined from the following variable: albumin, creatinine, fasting glucose, CRP, lymphocyte count, red cell size, alkaline phosphates, leukocyte count.

CONTACTS AND LOCATIONS:
Overall Officials: David JACOBI, PU-PH, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided